CLINICAL TRIAL: NCT03364309
Title: A Multicenter Study With a Randomized, Double-Blind, Placebo-Controlled Induction Dosing Period Followed by a Randomized Maintenance Dosing Period to Evaluate the Efficacy and Safety of LY2439821 in Chinese Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Study of Ixekizumab (LY2439821) in Chinese Participants With Moderate-to-Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14438; I1F-MC-RHBH (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-11-09; First posted 2017-12-06 (Actual); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06-01

CONDITIONS: Plaque Psoriasis
Keywords: plaque psoriasis; ixekizumab; skin condition; skin disease; itching; psoriasis vulgaris; immune-mediated systemic disease; skin lesions; scaly patches; papules
MeSH Terms: conditions — Skin Diseases; Pruritus | interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ixekizumab 80mg Q4W (Experimental): Participants received starting dose of 160 milligrams (mg) Ixekizumab at week 0 followed by 80mg Ixekizumab once every four weeks (Q4W) by subcutaneous injection during induction period.
  Interventions: Drug: Ixekizumab
- Ixekizumab 80mg Q2W (Experimental): Participants received starting dose of 160mg Ixekizumab at week 0 followed by 80mg Ixekizumab once every two weeks (Q2W) by subcutaneous injection during induction period.
  Interventions: Drug: Ixekizumab; Drug: Placebo
- Placebo (Placebo Comparator): Participants received placebo every two weeks (Q2W) by subcutaneous (SC)injection during induction period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821
  Arms: Ixekizumab 80mg Q2W; Ixekizumab 80mg Q4W
Drug: Placebo — Administered SC
  Arms: Ixekizumab 80mg Q2W; Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of the study drug ixekizumab in Chinese participants with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
Study I1F-MC-RHBH is a phase 3, multicenter, randomized, double-blind, placebo controlled, parallel-group study examining the effect of 2 dose regimens of ixekizumab versus placebo in participants with moderate-to-severe plaque psoriasis (Ps) during an induction dosing period with dosing for 12 weeks and the primary endpoint measured at 12 weeks, followed by a randomized, 48-week maintenance dosing period. During the maintenance dosing period, the study will evaluate the maintenance of response/remission, as well as relapse or rebound following treatment withdrawal, and response to retreatment following relapse.

ELIGIBILITY:
Inclusion Criteria:

* Present with chronic plaque Ps based on a confirmed diagnosis of chronic Ps vulgaris for at least 6 months prior to baseline.
* Have ≥10% BSA involvement at screening and baseline.
* Have both an sPGA score ≥3 and PASI score ≥12 at screening and baseline.
* Are candidates for phototherapy and/or systemic therapy.

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and/or guttate psoriasis) at screening or baseline.
* Drug-induced psoriasis.
* Ongoing use of prohibited treatments.
* Have previously completed or withdrawn from this study, or have previously exposed to ixekizumab or any other biologic drug directly targeting interleukin-17 (IL-17) (such as secukinumab) or the IL-17 receptor.
* Have concurrent or recent use of any biologic agent within washout periods or <5 half-lives prior to baseline, whichever is longer.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- China (17):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Guangdong Province People's Hospital, Guangzhou, Guangdong
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - YanCheng First People's Hospital, Yancheng, Jiangsu
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Nanjing
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Second Affiliate Hospital of Zhejiang Medical University, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Beijing Chao Yang Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University, Shanghai
  - Shanghai Dermatology Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Gao X, Pan W, Zheng M, Li F, Dong X, Lv D, Guo Z, Li J, Wang X, Geng S. Efficacy and Safety Analysis in Chinese Patients with Moderate-to-Severe Psoriasis from a Phase 3 Trial: Impact of Treatment Withdrawal and Retreatment of Ixekizumab. Adv Ther. 2025 Jan;42(1):334-347. doi: 10.1007/s12325-024-03030-5. Epub 2024 Nov 13. PMID 39535685
- [Derived] Li X, Ding Y, Zhang C, Lu Y, Li F, Pan W, Guo S, Li J, Zhao B, Zheng J. Efficacy of Ixekizumab in Chinese Patients with Moderate-to-Severe Psoriasis and Special Body Area Involvement: Sub-analysis of a Randomized, Double-Blind, Multicenter Phase 3 Study. Adv Ther. 2025 Jan;42(1):146-163. doi: 10.1007/s12325-024-02976-w. Epub 2024 Sep 30. PMID 39347926

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Responders were defined as achieving an sPGA score of 0 or 1. Non-responders were defined as having an sPGA score of >1. Responders were monitored for relapse, relapse (loss of response) occurring after Week 12 (Visit 7) was defined as an sPGA score of ≥3. In Re-treatment (Maintenance) Period, participants who relapsed received continued treatment of ixekizumab 80 mg Q4W, regardless of their treatment assignment.
Pre-assignment Details: Induction Dosing Period: Week 0 (baseline) to Week 12. Maintenance Dosing Period and Re-treatment (Maintenance) Period: Week 12 to Week 60.
  Post-Treatment Follow-Up Period: Occurred from last treatment period visit or Early Termination Visit (ETV) up to a minimum of 12 weeks following that visit.
Groups:
- PBO-Induction Dosing Period: Participants received placebo (PBO) every two weeks (Q2W) by subcutaneous (SC) injection during induction period.
- IXE80Q4W-Induction Dosing Period: Participants received starting dose of 160 milligrams (mg) Ixekizumab (IXE) at week 0 followed by 80mg Ixekizumab once every four weeks (80Q4W) by subcutaneous injection during induction period
- IXE80Q2W-Induction Dosing Period: Participants received starting dose of 160mg Ixekizumab at week 0 followed by 80mg Ixekizumab once every two weeks (80Q2W) by subcutaneous injection during induction period
- IXE80Q4W(Res)/PBO-Maintenance Dosing Period: Participants who received Ixekizumab 80mg Q4W in induction period and classified as responders received placebo Q4W by SC injection in maintenance dosing period.
- IXE80Q4W(Res)/IXE80Q4W-Maintenance Dosing Period: Participants who received Ixekizumab 80mg Q4W in induction period and classified as responders received Ixekizumab 80mg Q4W by SC injection in maintenance dosing period.
- IXE80Q2W(Res)/PBO-Maintenance Dosing Period: Participants who received Ixekizumab 80mg Q2W in induction period and classified as responders received placebo Q4W by SC injection in maintenance dosing period.
- IXE80Q2W(Res)/IXE80Q4W-Maintenance Dosing Period: Participants who received Ixekizumab 80mg Q2W in induction period and classified as responders received Ixekizumab 80mg Q4W by SC injection in maintenance dosing period.
- PBO(Res)/PBO-Maintenance Dosing Period: Participants who received placebo in induction period and classified as responders received placebo Q4W by SC injection in maintenance dosing period.
- PBO(NonResp)/IXE80Q4W-Maintenance Dosing Period: Participants who received placebo in induction period and classified as Non-responders (NonResp) received Ixekizumab 80 mg Q4W by SC injection in maintenance dosing period.
- IXE80Q4W(NonResp)/IXE80Q4W-Maintenance Dosing Period: Participants who received Ixekizumab 80mg Q4W in induction period and classified as Non-responders received Ixekizumab 80mg Q4W by SC injection in maintenance dosing period.
- IXE80Q2W(NonResp)/IXE80Q4W-Maintenance Dosing Period: Participants who received Ixekizumab 80mg Q2W in induction period and classified as non-responders received Ixekizumab 80mg Q4W by SC injection in maintenance dosing period.
- PBO(Resp)/PBO-Re-treatment (Maintenance) Period: Participants who were classified as placebo responders and received PBO during maintenance dosing period and after relapse retreated with Ixekizumab 80mg Q4W by SC injection.
- IXE80Q4W(Resp)/PBO-Re-treatment (Maintenance) Period: Participants who were classified as Ixekizumab 80mg Q4W responders and received PBO during maintenance dosing period and after relapse retreated with Ixekizumab 80mg Q4W by SC injection.
- IXE80Q4W(Resp)/IXE80Q4W-Re-treatment (Maintenance) Period: Participants who were classified as Ixekizumab 80mg Q4W responders and received Ixekizumab 80mg Q4W during maintenance dosing period and after relapse received Ixekizumab 80mg Q4W by SC injection.
- IXE80Q2W(Resp)/PBO-Re-treatment (Maintenance) Period: Participants who were classified as Ixekizumab 80mg Q2W responders and received PBO during maintenance dosing period and after relapse retreated with Ixekizumab 80mg Q4W by SC injection.
- IXE80Q2W(Resp)/IXE80Q4W-Re-treatment (Maintenance) Period: Participants who were classified as Ixekizumab 80mg Q2W responders and received Ixekizumab 80mg Q4W during maintenance dosing period and after relapse received Ixekizumab 80mg Q4W by SC injection.
- PBO-Follow-up Period; IXE80Q4W-Follow-up Period; IXE80Q2W-Follow-up Period: Participants did not receive any intervention in post treatment follow-up period
Period: Induction Period
Arm/Group | PBO-Induction Dosing Period | IXE80Q4W-Induction Dosing Period | IXE80Q2W-Induction Dosing Period | IXE80Q4W(Res)/PBO-Maintenance Dosing Period | IXE80Q4W(Res)/IXE80Q4W-Maintenance Dosing Period | IXE80Q2W(Res)/PBO-Maintenance Dosing Period | IXE80Q2W(Res)/IXE80Q4W-Maintenance Dosing Period | PBO(Res)/PBO-Maintenance Dosing Period | PBO(NonResp)/IXE80Q4W-Maintenance Dosing Period | IXE80Q4W(NonResp)/IXE80Q4W-Maintenance Dosing Period | IXE80Q2W(NonResp)/IXE80Q4W-Maintenance Dosing Period | PBO(Resp)/PBO-Re-treatment (Maintenance) Period | IXE80Q4W(Resp)/PBO-Re-treatment (Maintenance) Period | IXE80Q4W(Resp)/IXE80Q4W-Re-treatment (Maintenance) Period | IXE80Q2W(Resp)/PBO-Re-treatment (Maintenance) Period | IXE80Q2W(Resp)/IXE80Q4W-Re-treatment (Maintenance) Period | PBO-Follow-up Period | IXE80Q4W-Follow-up Period | IXE80Q2W-Follow-up Period
Started | 88 | 174 | 176 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 88 | 174 | 176 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 82 | 170 | 175 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Period
Arm/Group | PBO-Induction Dosing Period | IXE80Q4W-Induction Dosing Period | IXE80Q2W-Induction Dosing Period | IXE80Q4W(Res)/PBO-Maintenance Dosing Period | IXE80Q4W(Res)/IXE80Q4W-Maintenance Dosing Period | IXE80Q2W(Res)/PBO-Maintenance Dosing Period | IXE80Q2W(Res)/IXE80Q4W-Maintenance Dosing Period | PBO(Res)/PBO-Maintenance Dosing Period | PBO(NonResp)/IXE80Q4W-Maintenance Dosing Period | IXE80Q4W(NonResp)/IXE80Q4W-Maintenance Dosing Period | IXE80Q2W(NonResp)/IXE80Q4W-Maintenance Dosing Period | PBO(Resp)/PBO-Re-treatment (Maintenance) Period | IXE80Q4W(Resp)/PBO-Re-treatment (Maintenance) Period | IXE80Q4W(Resp)/IXE80Q4W-Re-treatment (Maintenance) Period | IXE80Q2W(Resp)/PBO-Re-treatment (Maintenance) Period | IXE80Q2W(Resp)/IXE80Q4W-Re-treatment (Maintenance) Period | PBO-Follow-up Period | IXE80Q4W-Follow-up Period | IXE80Q2W-Follow-up Period
Started | 0 (This period is to report Maintenance Period participants.) | 0 (This period is to report Maintenance Period participants.) | 0 (This period is to report Maintenance Period participants.) | 47 (This period is to report Maintenance Period participants.) | 92 (This period is to report Maintenance Period participants.) | 50 (This period is to report Maintenance Period participants.) | 100 (This period is to report Maintenance Period participants.) | 3 (This period is to report Maintenance Period participants.) | 79 (This period is to report Maintenance Period participants.) | 31 (This period is to report Maintenance Period participants.) | 23 (This period is to report Maintenance Period participants.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 0 | 0 | 0 | 47 | 92 | 50 | 100 | 3 | 79 | 31 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 3 | 80 | 4 | 84 | 1 | 73 | 27 | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 44 | 12 | 46 | 16 | 2 | 6 | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 3 | 1 | 3 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Relapsed | 0 | 0 | 0 | 43 | 7 | 45 | 10 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Miscellaneous | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Re-treatment (Maintenance) Period
Arm/Group | PBO-Induction Dosing Period | IXE80Q4W-Induction Dosing Period | IXE80Q2W-Induction Dosing Period | IXE80Q4W(Res)/PBO-Maintenance Dosing Period | IXE80Q4W(Res)/IXE80Q4W-Maintenance Dosing Period | IXE80Q2W(Res)/PBO-Maintenance Dosing Period | IXE80Q2W(Res)/IXE80Q4W-Maintenance Dosing Period | PBO(Res)/PBO-Maintenance Dosing Period | PBO(NonResp)/IXE80Q4W-Maintenance Dosing Period | IXE80Q4W(NonResp)/IXE80Q4W-Maintenance Dosing Period | IXE80Q2W(NonResp)/IXE80Q4W-Maintenance Dosing Period | PBO(Resp)/PBO-Re-treatment (Maintenance) Period | IXE80Q4W(Resp)/PBO-Re-treatment (Maintenance) Period | IXE80Q4W(Resp)/IXE80Q4W-Re-treatment (Maintenance) Period | IXE80Q2W(Resp)/PBO-Re-treatment (Maintenance) Period | IXE80Q2W(Resp)/IXE80Q4W-Re-treatment (Maintenance) Period | PBO-Follow-up Period | IXE80Q4W-Follow-up Period | IXE80Q2W-Follow-up Period
Started | 0 | 0 | 0 | 0 (This period is to report for Re-treatment (Maintenance) Period.) | 0 (This period is to report for Re-treatment (Maintenance) Period.) | 0 (This period is to report for Re-treatment (Maintenance) Period.) | 0 (This period is to report for Re-treatment (Maintenance) Period.) | 0 (This period is to report for Re-treatment (Maintenance) Period.) | 0 (This period is to report for Re-treatment (Maintenance) Period.) | 0 (This period is to report for Re-treatment (Maintenance) Period.) | 0 (This period is to report for Re-treatment (Maintenance) Period.) | 2 (This period is to report for Re-treatment (Maintenance) Period.) | 43 (This period is to report for Re-treatment (Maintenance) Period.) | 7 (This period is to report for Re-treatment (Maintenance) Period.) | 45 (This period is to report for Re-treatment (Maintenance) Period.) | 10 (This period is to report for Re-treatment (Maintenance) Period.) | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 42 | 6 | 43 | 8 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Relapse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Period: Post-Treatment Followup Period
Arm/Group | PBO-Induction Dosing Period | IXE80Q4W-Induction Dosing Period | IXE80Q2W-Induction Dosing Period | IXE80Q4W(Res)/PBO-Maintenance Dosing Period | IXE80Q4W(Res)/IXE80Q4W-Maintenance Dosing Period | IXE80Q2W(Res)/PBO-Maintenance Dosing Period | IXE80Q2W(Res)/IXE80Q4W-Maintenance Dosing Period | PBO(Res)/PBO-Maintenance Dosing Period | PBO(NonResp)/IXE80Q4W-Maintenance Dosing Period | IXE80Q4W(NonResp)/IXE80Q4W-Maintenance Dosing Period | IXE80Q2W(NonResp)/IXE80Q4W-Maintenance Dosing Period | PBO(Resp)/PBO-Re-treatment (Maintenance) Period | IXE80Q4W(Resp)/PBO-Re-treatment (Maintenance) Period | IXE80Q4W(Resp)/IXE80Q4W-Re-treatment (Maintenance) Period | IXE80Q2W(Resp)/PBO-Re-treatment (Maintenance) Period | IXE80Q2W(Resp)/IXE80Q4W-Re-treatment (Maintenance) Period | PBO-Follow-up Period | IXE80Q4W-Follow-up Period | IXE80Q2W-Follow-up Period
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (This period is to report for Follow-up Period participants.) | 0 (This period is to report for Follow-up Period participants.) | 0 (This period is to report for Follow-up Period participants.) | 0 (This period is to report for Follow-up Period participants.) | 0 (This period is to report for Follow-up Period participants.) | 11 (This period is to report for Follow-up Period participants.) | 375 (This period is to report for Follow-up Period participants.) | 2 (This period is to report for Follow-up Period participants.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 344 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 31 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 19 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Miscellaneous | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Ixekizumab 80mg Q2W | Total
Number analyzed (Participants) | 88 | 174 | 176 | 438
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (12.38) | 41.2 (11.59) | 39.2 (10.53) | 40.5 (11.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 45 | 34 | 103
  Male | 64 | 129 | 142 | 335
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 88 | 174 | 176 | 438
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 88 | 174 | 176 | 438

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Static Physician Global Assessment (sPGA) Score of Clear (0) or Minimal (1) With at Least a 2 Point Improvement
Description: The sPGA is the physician's determination of the participant's Ps lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participants Ps were assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe). An sPGA responder was defined as having a post-baseline sPGA score of "0" or "1" with at least a 2-point improvement from baseline.
Time Frame: Week 12
Population: All randomized participants with baseline sPGA >=3 & received at least 1 dose of study drug and had a post-baseline measurement for sPGA. Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 88 | 174 | 176
Percentage of participants | 3.4 [0.0 to 7.2] | 79.9 [73.9 to 85.8] | 86.4 [81.3 to 91.4]
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 99.99, 95% CI 2-sided [33.57 to 99.99]
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 99.99, 95% CI 2-sided [52.49 to 99.99]

2. Primary Outcome: Percentage of Participants Achieving a ≥75% Improvement in Psoriasis Area and Severity Index (PASI 75)
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored by itself and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease).
Time Frame: Week 12
Population: All randomized participants who received at least 1 dose of study drug and had a post-baseline measurement for PASI 75. Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 88 | 174 | 176
Percentage of participants | 8.0 [2.3 to 13.6] | 87.4 [82.4 to 92.3] | 93.8 [90.2 to 97.3]
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 79.95, 95% CI 2-sided [32.76 to 99.99]
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 99.99, 95% CI 2-sided [64.87 to 99.99]

3. Secondary Outcome: Percentage of Participants Achieving a Static Physician Global Assessment (sPGA) Score of Clear (0) (Remission)
Description: The sPGA is the physician's determination of the participant's Ps lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participants Ps were assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe). An sPGA assessed as 0, indicates complete resolution of plaque Ps.
Time Frame: Week 12
Population: All randomized participants who received at least 1 dose of study drug and had a post-baseline measurement for sPGA (0). Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 88 | 174 | 176
Percentage of participants | 0.0 [0.0 to 0.0] | 35.6 [28.5 to 42.7] | 36.4 [29.3 to 43.5]

4. Secondary Outcome: Percentage of Participants Achieving a ≥90% Improvement in Psoriasis Area and Severity Index (PASI 90)
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored by itself and the scores were then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease).
Time Frame: Week 12
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post-baseline measurement for PASI 90. Participants who did not meet the clinical response criteria or had missing data were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 88 | 174 | 176
Percentage of participants | 2.3 [0.0 to 5.4] | 75.9 [69.5 to 82.2] | 82.4 [76.8 to 88.0]
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 99.99, 95% CI 2-sided [31.88 to 99.99]
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 99.99, 95% CI 2-sided [46.96 to 99.99]

5. Secondary Outcome: Percentage of Participants Achieving a 100% Improvement in Psoriasis Area and Severity Index (PASI 100)
Description: as for outcome 4
Time Frame: Week 12
Population: All randomized participants who received at least 1 dose of study drug and had a post-baseline measurement for PASI 100. Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 88 | 174 | 176
Percentage of participants | 0.0 [0.0 to 0.0] | 29.3 [22.5 to 36.1] | 33.0 [26.0 to 39.9]

6. Secondary Outcome: Percentage of Participants Achieving an Itch Numeric Rating Scale (NRS) ≥4 Point Reduction From Baseline for Participants Who Had Baseline Itch NRS ≥4
Description: The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 (no itch) and 10 (worst itch imaginable). Overall severity of a participant's itching from Ps is indicated by circling the number that best describes the worst level of itching in the past 24 hours.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had baseline who had baseline Itch NRS ≥4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 62 | 128 | 125
percentage of participants | 8.1 [1.3 to 14.8] | 76.6 [69.2 to 83.9] | 78.4 [71.2 to 85.6]
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 37.24, 95% CI 2-sided [13.68 to 99.99]
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 41.38, 95% CI 2-sided [15.09 to 99.99]

7. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score
Description: The DLQI is a simple, participant-administered, 10 question, validated, quality-of-life questionnaire that covers 6 domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include "not at all," "a lot," and "very much," with corresponding scores of 1, 2, and 3, respectively, and unanswered ("not relevant") responses scored as "0." Totals range from 0 to 30 (less to more impairment). A score of 0 or 1 indicates no impact of disease on a participants quality of life.
  Least Square Mean (LS Mean) was calculated using Mixed Model Repeated Measures (MMRM) model includes treatment, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had baseline and post baseline DLQI total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 82 | 170 | 175
units on a scale | 0.92 (0.495) | -8.60 (0.346) | -8.86 (0.343)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -9.52, 95% CI 2-sided [-10.71 to -8.33], Standard Error of Mean 0.604
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -9.78, 95% CI 2-sided [-10.96 to -8.59], Standard Error of Mean 0.603

8. Secondary Outcome: Change From Baseline in Nail Psoriasis Severity Index (NAPSI) Score in Participants With Baseline Fingernail Involvement
Description: NAPSI is a numeric, reproducible, objective tool for evaluation of fingernail(fn) Ps. This scale is used to evaluate severity of fn bed Ps & fn matrix Ps by area of involvement in the fn unit. fn is divided with imaginary horizontal & longitudinal lines into quadrants. Each fn is given a score for fn bed Ps 0(none) to 4(Ps in 4 quadrants of the fn) & fn matrix Ps 0(none) to 4(Ps in 4 quadrants in matrix), depending on presence (score of 1) or absence (score of 0) of any of the features of fn bed or matrix Ps in each quadrant.NAPSI score of a fn is sum of scores in fn bed & fn matrix from each quadrant (maximum of 8). Each fn is evaluated, then the sum of all fn equals the total NAPSI score with a range from range 0 to 80. Higher scores indicate more severe ps. LS Mean was calculated using MMRM model includes treatment, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had baseline fingernail involvement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 66 | 132 | 130
units on a scale | -1.26 (1.365) | -11.35 (0.967) | -10.07 (0.974)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -10.09, 95% CI 2-sided [-13.38 to -6.79], Standard Error of Mean 1.673
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -8.81, 95% CI 2-sided [-12.11 to -5.51], Standard Error of Mean 1.677

9. Secondary Outcome: Change From Baseline in Percent of Body Surface Area (BSA) Involvement of Psoriasis
Description: The percentage involvement of psoriasis on each participant's body surface area was assessed by the investigator on a scale from 0% (no involvement) to 100% (full involvement), in which 1% corresponds to the size of the participant's hand including palm, fingers and thumb.
  LS Mean was calculated using MMRM model includes treatment, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had postbaseline BSA involvement.
Measure: Least Squares Mean (Standard Error); unit: Percent of BSA
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 82 | 170 | 175
Percent of BSA | -0.36 (1.660) | -35.32 (1.157) | -36.70 (1.146)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -34.96, 95% CI 2-sided [-38.94 to -30.98], Standard Error of Mean 2.023
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -36.34, 95% CI 2-sided [-40.30 to -32.37], Standard Error of Mean 2.018

10. Secondary Outcome: Change From Baseline in Psoriasis Scalp Severity Index (PSSI) Score in Participants With Baseline Scalp Involvement
Description: The PSSI is a physician assessment of erythema, induration and desquamation and percent of scalp that is covered with a scores range from 0 (none) to 4 (very severe). The composite score is derived from the sum of scores for erythema, induration, and desquamation multiplied by the score recorded for the extent of the scalp area involved, 1 (<10%) to 6 (90%-100%) with a total score ranging from 0 (less severity) to 72 (more severity). LS Mean was calculated using MMRM model includes treatment, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had baseline scalp involvement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 78 | 166 | 171
units on a scale | -1.59 (0.787) | -18.33 (0.544) | -19.52 (0.539)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -16.74, 95% CI 2-sided [-18.62 to -14.86], Standard Error of Mean 0.957
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -17.93, 95% CI 2-sided [-19.80 to -16.05], Standard Error of Mean 0.954

11. Secondary Outcome: Change From Baseline in Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS) Score
Description: The SF-36 is a participant-reported outcome measure evaluating participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. Items from 8 domains contribute to the PCS. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health. LS Mean was calculated using MMRM model includes treatment, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had post baseline SF-36 PCS score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 82 | 170 | 175
units on a scale | -1.812 (0.5492) | 4.417 (0.3815) | 4.724 (0.3766)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = 6.228, 95% CI 2-sided [4.915 to 7.541], Standard Error of Mean 0.6681
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = 6.536, 95% CI 2-sided [5.225 to 7.847], Standard Error of Mean 0.6668

12. Secondary Outcome: Change From Baseline in Medical Outcomes Study SF-36 Mental Component Summary (MCS) Score
Description: as for outcome 11
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had post baseline SF-36 MCS score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 82 | 170 | 175
units on a scale | -1.233 (0.7798) | 3.960 (0.5414) | 4.129 (0.5342)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = 5.193, 95% CI 2-sided [3.328 to 7.058], Standard Error of Mean 0.9489
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = 5.362, 95% CI 2-sided [3.503 to 7.222], Standard Error of Mean 0.9460

13. Secondary Outcome: Change From Baseline on Patient Global Assessment of Disease Severity
Description: The Patient Global Assessment of Disease Severity is a single-item participant-reported outcome measure on which participants are asked to rate the severity of their psoriasis "today" from 0 (Clear) = no psoriasis, to 5 (Severe) = the worst their psoriasis has ever been.
  LS Mean was calculated using MMRM model includes treatment, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had postbaseline patient global assessment score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 82 | 170 | 175
units on a scale | -0.5 (0.12) | -3.1 (0.08) | -3.1 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -2.6, 95% CI 2-sided [-2.9 to -2.4], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -2.6, 95% CI 2-sided [-2.9 to -2.3], Standard Error of Mean 0.15

14. Secondary Outcome: Change From Baseline in Palmoplantar PASI (PPASI) in Participants With Baseline Palmoplantar Involvement
Description: The Palmoplantar PASI is a composite score derived from the sum scores for erythema, induration, and desquamation multiplied by a score for the extent of palm and sole area involvement, ranging from 0 (no Ps) to 72. (the most severe disease) The PPASI was only assessed if participants have palmoplantar psoriasis at baseline. LS Mean was calculated using MMRM model includes treatment, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had baseline palmoplantar psoriasis involvement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 26 | 41 | 51
units on a scale | -2.99 (0.861) | -6.34 (0.688) | -7.78 (0.626)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p = 0.003, Mixed Models Analysis; LSMean Difference = -3.35, 95% CI 2-sided [-5.56 to -1.15], Standard Error of Mean 1.110
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -4.79, 95% CI 2-sided [-6.90 to -2.67], Standard Error of Mean 1.064

15. Secondary Outcome: Change From Baseline on the Joint Pain Visual Analog Scale (VAS)
Description: The Joint Pain VAS is a participant-administered scale designed to measure current joint pain from PsA using a 100-mm horizontal VAS. Overall severity of a participant's joint pain from PsA is indicated by placing a single mark on the horizontal scale (0 = none; 100 = as severe as you can imagine). LS Mean was calculated using MMRM model includes treatment, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had baseline psoriatic arthritis.
Measure: Least Squares Mean (Standard Error); unit: millimeter (mm)
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 3 | 8 | 12
millimeter (mm) | -12.2 (9.64) | -39.6 (5.48) | -37.4 (4.75)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p = 0.022, Mixed Models Analysis; LSMean Difference = -27.4, 95% CI 2-sided [-50.5 to -4.3], Standard Error of Mean 11.07
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80mg Q2W; Test type: Superiority; p = 0.031, Mixed Models Analysis; LSMean Difference = -25.2, 95% CI 2-sided [-47.8 to -2.5], Standard Error of Mean 10.87

16. Secondary Outcome: Percentage of Participants With Anti-Ixekizumab Antibodies
Description: Percentage was calculated based on the number of evaluable participants and was calculated by number of participants with treatment-emergent positive anti-ixekizumab antibodies / number of evaluable participants * 100%.
Time Frame: Baseline through Week 12
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Ixekizumab 80mg Q2W
Number analyzed (Participants) | 88 | 174 | 176
percentage of participants | 0 | 19 | 12.5

ADVERSE EVENTS:
Time Frame: Up to 72 weeks
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- PBO-Induction Dosing Period: Participants received placebo every two weeks (Q2W) by subcutaneous (SC)injection during induction period.
- IXE80Q4W-Induction Dosing Period: Participants received starting dose of 160 milligrams (mg) Ixekizumab at week 0 followed by 80mg Ixekizumab once every four weeks (Q4W) by subcutaneous injection during induction period
- IXE80Q2W-Induction Dosing Period: Participants received starting dose of 160mg Ixekizumab at week 0 followed by 80mg Ixekizumab once every two weeks (Q2W) by subcutaneous injection during induction period
- PBO(NonResp)/IXE80Q4W-Maintenance Dosing Period: Participants who received placebo in induction period and classified as Non-responders received Ixekizumab 80mg Q4W by SC injection in maintenance dosing period.
Arm/Group | PBO-Induction Dosing Period | IXE80Q4W-Induction Dosing Period | IXE80Q2W-Induction Dosing Period | IXE80Q4W(Res)/PBO-Maintenance Dosing Period | IXE80Q4W(Res)/IXE80Q4W-Maintenance Dosing Period | IXE80Q2W(Res)/PBO-Maintenance Dosing Period | IXE80Q2W(Res)/IXE80Q4W-Maintenance Dosing Period | PBO(Res)/PBO-Maintenance Dosing Period | PBO(NonResp)/IXE80Q4W-Maintenance Dosing Period | IXE80Q4W(NonResp)/IXE80Q4W-Maintenance Dosing Period | IXE80Q2W(NonResp)/IXE80Q4W-Maintenance Dosing Period | PBO(Resp)/PBO-Re-treatment (Maintenance) Period | IXE80Q4W(Resp)/PBO-Re-treatment (Maintenance) Period | IXE80Q4W(Resp)/IXE80Q4W-Re-treatment (Maintenance) Period | IXE80Q2W(Resp)/PBO-Re-treatment (Maintenance) Period | IXE80Q2W(Resp)/IXE80Q4W-Re-treatment (Maintenance) Period | PBO-Follow-up Period | IXE80Q4W-Follow-up Period | IXE80Q2W-Follow-up Period
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/174 | 0/176 | 0/47 | 0/92 | 0/50 | 0/100 | 0/3 | 1/79 | 0/31 | 0/23 | 0/2 | 0/43 | 0/7 | 0/45 | 0/10 | 0/11 | 0/375 | 0/2
Serious Adverse Events (participants affected / at risk) | 3/88 | 2/174 | 1/176 | 1/47 | 5/92 | 1/50 | 2/100 | 1/3 | 5/79 | 0/31 | 1/23 | 0/2 | 1/43 | 0/7 | 2/45 | 0/10 | 0/11 | 7/375 | 0/2
Other Adverse Events (participants affected / at risk) | 25/88 | 89/174 | 97/176 | 24/47 | 68/92 | 22/50 | 66/100 | 1/3 | 58/79 | 22/31 | 14/23 | 1/2 | 24/43 | 4/7 | 27/45 | 5/10 | 0/11 | 27/375 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | PBO-Induction Dosing Period (N=88) | IXE80Q4W-Induction Dosing Period (N=174) | IXE80Q2W-Induction Dosing Period (N=176) | IXE80Q4W(Res)/PBO-Maintenance Dosing Period (N=47) | IXE80Q4W(Res)/IXE80Q4W-Maintenance Dosing Period (N=92) | IXE80Q2W(Res)/PBO-Maintenance Dosing Period (N=50) | IXE80Q2W(Res)/IXE80Q4W-Maintenance Dosing Period (N=100) | PBO(Res)/PBO-Maintenance Dosing Period (N=3) | PBO(NonResp)/IXE80Q4W-Maintenance Dosing Period (N=79) | IXE80Q4W(NonResp)/IXE80Q4W-Maintenance Dosing Period (N=31) | IXE80Q2W(NonResp)/IXE80Q4W-Maintenance Dosing Period (N=23) | PBO(Resp)/PBO-Re-treatment (Maintenance) Period (N=2) | IXE80Q4W(Resp)/PBO-Re-treatment (Maintenance) Period (N=43) | IXE80Q4W(Resp)/IXE80Q4W-Re-treatment (Maintenance) Period (N=7) | IXE80Q2W(Resp)/PBO-Re-treatment (Maintenance) Period (N=45) | IXE80Q2W(Resp)/IXE80Q4W-Re-treatment (Maintenance) Period (N=10) | PBO-Follow-up Period (N=11) | IXE80Q4W-Follow-up Period (N=375) | IXE80Q2W-Follow-up Period (N=2)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/24 (0) | 0/45 (0) | 0/34 (0) | 0/10 (0) | 1/27 (1) | 0/14 (0) | 0/15 (0) | 0/1 (0) | 0/21 (0) | 0/5 (0) | 0/3 (0) | 0/1 (0) | 0/10 (0) | 0/3 (0) | 0/12 (0) | 0/1 (0) | 0/3 (0) | 0/84 (0) | 0/1 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrosalpinx (Reproductive system and breast disorders) | 0/24 (0) | 0/45 (0) | 0/34 (0) | 0/10 (0) | 0/27 (0) | 0/14 (0) | 0/15 (0) | 1/1 (1) | 0/21 (0) | 0/5 (0) | 0/3 (0) | 0/1 (0) | 0/10 (0) | 0/3 (0) | 0/12 (0) | 0/1 (0) | 0/3 (0) | 0/84 (0) | 0/1 (0)
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PBO-Induction Dosing Period (N=88) | IXE80Q4W-Induction Dosing Period (N=174) | IXE80Q2W-Induction Dosing Period (N=176) | IXE80Q4W(Res)/PBO-Maintenance Dosing Period (N=47) | IXE80Q4W(Res)/IXE80Q4W-Maintenance Dosing Period (N=92) | IXE80Q2W(Res)/PBO-Maintenance Dosing Period (N=50) | IXE80Q2W(Res)/IXE80Q4W-Maintenance Dosing Period (N=100) | PBO(Res)/PBO-Maintenance Dosing Period (N=3) | PBO(NonResp)/IXE80Q4W-Maintenance Dosing Period (N=79) | IXE80Q4W(NonResp)/IXE80Q4W-Maintenance Dosing Period (N=31) | IXE80Q2W(NonResp)/IXE80Q4W-Maintenance Dosing Period (N=23) | PBO(Resp)/PBO-Re-treatment (Maintenance) Period (N=2) | IXE80Q4W(Resp)/PBO-Re-treatment (Maintenance) Period (N=43) | IXE80Q4W(Resp)/IXE80Q4W-Re-treatment (Maintenance) Period (N=7) | IXE80Q2W(Resp)/PBO-Re-treatment (Maintenance) Period (N=45) | IXE80Q2W(Resp)/IXE80Q4W-Re-treatment (Maintenance) Period (N=10) | PBO-Follow-up Period (N=11) | IXE80Q4W-Follow-up Period (N=375) | IXE80Q2W-Follow-up Period (N=2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous opacities (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site hypersensitivity (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 13 (18) | 19 (43) | 0 (0) | 17 (62) | 0 (0) | 17 (64) | 0 (0) | 8 (40) | 3 (6) | 2 (12) | 0 (0) | 3 (5) | 1 (2) | 5 (20) | 1 (10) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (4) | 0 (0) | 3 (19) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 1 (5) | 2 (13) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 10 (10) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 0 (0) | 4 (5) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 6 (7) | 0 (0) | 4 (4) | 2 (5) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 4 (5) | 8 (10) | 2 (3) | 6 (7) | 2 (4) | 4 (4) | 0 (0) | 3 (6) | 1 (1) | 3 (4) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 5 (7) | 4 (4) | 0 (0) | 5 (5) | 1 (1) | 6 (6) | 0 (0) | 9 (9) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 9 (9) | 9 (9) | 3 (3) | 11 (12) | 3 (3) | 10 (11) | 0 (0) | 6 (11) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (10) | 25 (27) | 28 (34) | 7 (8) | 25 (35) | 6 (6) | 31 (42) | 0 (0) | 22 (24) | 8 (12) | 3 (4) | 1 (1) | 7 (8) | 2 (2) | 9 (11) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 2 (4) | 4 (4) | 3 (3) | 2 (2) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 2 (3) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Blood immunoglobulin a increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count abnormal (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 3 (3) | 5 (5) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine ketone body present (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 6 (6) | 3 (3) | 2 (2) | 4 (4) | 0 (0) | 3 (4) | 0 (0) | 6 (6) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 3 (4) | 1 (1) | 5 (7) | 1 (1) | 5 (6) | 0 (0) | 3 (5) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 2 (2) | 2 (2) | 2 (2) | 2 (3) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 3 (4) | 0 (0) | 8 (9) | 2 (3) | 5 (5) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 5 (5) | 4 (8) | 2 (2) | 5 (6) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (5) | 1 (2) | 8 (8) | 0 (0) | 6 (8) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (11) | 8 (9) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (7) | 10 (10) | 1 (1) | 4 (5) | 0 (0) | 7 (10) | 0 (0) | 9 (12) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 5 (5) | 4 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT03364309/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT03364309/SAP_001.pdf